CLINICAL TRIAL: NCT00290420
Title: Prevention of P. Vivax Malaria During Pregnancy: Effects on Mother and Child Health in Santa Cruz, Bolivia. Open, Multicentric, Randomized Clinical Trial, Comparing Prophylaxis Once a Week to Malaria Attack Treatment, Both by Chloroquine.
Brief Title: Prevention of P. Vivax Malaria During Pregnancy in Bolivia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: important delays and malaria season missed, due to political changes
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Instituto Nacional de Laboratorios de Salud (INLASA) (Unknown); Pan American Health Organization (Other); Ministry of Health, Bolivia (Other Government)
Responsible Party: Principal Investigator, Bernadette Murgue, administrative responsible for IRD, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRD/Prevmal/Bol/06
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Malaria
Keywords: malaria; Plasmodium vivax; pregnancy; chemoprophylaxis
MeSH Terms: conditions — Malaria; Malaria, Vivax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine profilaxis (Experimental): Prevention: chloroquine profilaxis
  Prevention of malaria attacks with chloroquine profilaxis taken once a week
  Interventions: Drug: Chloroquine profilaxis
- No prevention (No Intervention): Treatment of malaria attack with chloroquine when they occur

INTERVENTIONS:
Drug: Chloroquine profilaxis — Prevention:
  Give a profilaxis with chloroquine once a week to prevent Plasmodium vivax malaria attacks and to prevent harmfull effect on birth outcomes
  Other Names: prevention of plasmodium vivax malaria harmfull effects on birth outcomes
  Arms: Chloroquine profilaxis

SUMMARY:
The purpose of this study is to determine which, between weekly prophylaxis or malaria attack treatment, both by chloroquine, is the most appropriate way to protect women and foetus from P. vivax malaria infection during pregnancy.

DETAILED DESCRIPTION:
It has been demonstrated that malaria is responsible for anaemia during pregnancy and reduces birth weight among newborns. In Bolivia, malaria is mostly caused by P. vivax. Maternal and foetal consequences of P. vivax infections have been poorly investigated until now, over all in South America. In fact, recommendations for the protection of pregnant women from malaria in Bolivia have not been clearly established. Prophylaxis by chloroquine is still recommended in other continents than Africa, mainly because chloroquine resistances are still uncommon in P. vivax species. The alternative way to protect women during pregnancy is to treat malaria attacks during antenatal visits. For this purpose, we will realize a study in order to assess the most appropriate way to protect women and foetus from malaria infection, i.e. weekly prophylaxis or mild malaria attack treatment, both by chloroquine. By realizing a randomized and multicentric clinical trial on 800 women in each group, we will compare the impact on maternal malaria attack incidence rates, on proportions of mothers with anaemia, on low-birth weight and on positive parasitaemias during pregnancy and at delivery, of weekly prophylaxis and mild malaria attack diagnosis and treatment. The study will be undertaken during 18 months in the region of Santa Cruz and will give important information to the Bolivian Ministry of Health for establishing national recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 4 to 36 weeks of gestation
* Intention to deliver at the maternity clinics
* Residence near the maternity clinics
* Written informed consent (parents or tutors if aged<18 years)

Exclusion Criteria:

* Pregnancy prior to 4 weeks or after 36 weeks of gestation
* Allergy to chloroquine
* Clinical signs of hepatic or renal alteration
* Inability to take drugs by oral route
* Presence of effective uterine contractions

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Estimated); Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of women presenting a malaria attack during pregnancy | two years

SECONDARY OUTCOMES:
proportions of mothers with placental plasmodial infection | 2 years
proportions of mothers with moderate to severe anaemia (<8g/dl) at delivery | 2 years
maternal haemoglobin rate at delivery | 2 years
proportions of women with parasitaemia during pregnancy and at delivery | 2 years
mean parasites densities of women with parasitaemia during pregnancy and at delivery | 2 years
proportions of children with low birthweight (<2,500 grams) | 2 years
mean birthweight | 2 years
proportions of preterm deliveries | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michel Cot, MD-PhD, Study Director — Institut de Recherche pour le Developpement; Laurent Brutus, MD-MSc, Study Director — Institut de Recherche pour le Développement, IRD, Bolivia; Agnès Le Port, MSc, Principal Investigator — Institut de Recherche pour le Développement, IRD, Bolivia